CLINICAL TRIAL: NCT02251210
Title: Three Month, Randomised, Double-blind, Double-dummy, Placebo-controlled, Multiple Dose-range Study of the Efficacy and Safety of BIIL 284 BS (5, 25 and 75 mg p.o. Once Daily) in Adult Patients With Active Rheumatoid Arthritis
Brief Title: Efficacy and Safety of BIIL 284 BS in Adult Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.27
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — amelubant

ARMS (4):
- BIIL 284 BS low dose (Experimental)
  Interventions: Drug: BIIL 284 BS low dose
- BIIL 284 BS medium dose (Experimental)
  Interventions: Drug: BIIL 284 BS medium dose
- BIIL 284 BS high dose (Experimental)
  Interventions: Drug: BIIL 284 BS high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS low dose
  Arms: BIIL 284 BS low dose
Drug: BIIL 284 BS medium dose
  Arms: BIIL 284 BS medium dose
Drug: BIIL 284 BS high dose
  Arms: BIIL 284 BS high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate efficacy and safety of 3 doses of BIIL 284 BS in active rheumatoid arthritis (RA) and determine the dose with most positive efficacy / safety ratio. Pharmacokinetic profile will be also obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients of >=18 and <= 70 years of age
* Patients suffering from rheumatoid arthritis as defined by the American Rheumatism Association (ARA) criteria revised 1987 and date of diagnosis >= 6 months. At least 4 of the following 7 criteria must be present:

  * Morning stiffness in and around the joints lasting at least 1 hour before maximal improvement for at least 6 weeks
  * Arthritis (soft tissue thickening or fluid - not bony overgrowth alone) of at least 3 joint areas for at least 6 weeks
  * Arthritis of hand joints (at least one area swollen in a wrist, metacarpophalangeal (MCP) or proximal interphalangeal (PIP) joint) for at least 6 weeks
  * Symmetrical arthritis (observed by a physician) with simultaneous involvement of the joints on both sides of the body for at least 6 weeks
  * Rheumatoid nodules (observed by a physician) over bony prominence or extensor surfaces or in juxta-articular regions
  * Serum rheumatoid factor positive
  * X-ray changes typical of rheumatoid arthritis (erosions or unequivocal bony decalcification localized in or most marked adjacent to the involved joints)
* Patients belonging to the RA functional class I, II or III
* Active RA as defined at visit 2 by:

  * Swollen joint count at least of 6 (of 28 joints examined) and
  * Tender joint count at least of 8 (of 28 joints examined) and
  * Patients must fulfil 2 out of the 3 following criteria:

    * Patient's assessment of pain (VAS) >= 40 mm
    * Investigator's global assessment of disease activity on a VAS >= 40 mm
    * ESR >= 28 mm/h or CRP >= 20 mg/L
* Patient's written informed consent obtained at Visit 1 (screening) before enrolment in the study

Exclusion Criteria:

* Patient presenting or having a history of inflammatory rheumatic disease other than RA (e.g.: mixed connective tissue disease, systemic lupus erythematosus, seronegative spondyloarthropathy)
* Patients who have failed to more than 3 different disease-modifying antirheumatic drug (DMARDs) therapies previously due to lack of efficacy (in case of combined therapy each DMARDs used is counted as one)
* Patients with any other disease that could interfere with the evaluation of efficacy and safety
* Patients in treatment with any DMARDs / slow-acting anti-rheumatic drug (SAARDs) during the periods specified:

  * 4 weeks before V2: Methotrexate, parenteral/oral gold, D-penicillamine, Sulphasalazine, antimalarials (e.g.:Chloroquine/Hydroxychloroquine), Azathioprine, Cyclosporine A, Alkylating agents (e.g.: Cyclophosphamide / Chlorambucil), Minocycline, Etanercept (Enbrel®), and Leflunomide (only if wash-out with Colestyramine has been done after leflunomide discontinuation)
  * 3 months before Visit 2: Leflunomide if no wash- out with colestyramine has been done after leflunomide discontinuation, Infliximab (Remicade®), any other biological compound.
* Patient in treatment with oral corticosteroids at a dose higher than 10 mg/day or 0.2 mg/Kg/day (prednisone equivalent) whichever is lower, during the 4 weeks prior to Visit 2, change in the treatment with oral corticosteroids during the 4 weeks prior to Visit 2 or intended change during the trial
* Patients in treatment with any parenteral (intravenous, intramuscular or intraarticular) treatment with corticosteroids during the 4 weeks prior to Visit 2 or their intended use during the trial.
* Change in treatment with non-steroidal anti-inflammatory drugs (NSAIDs) during the 2 weeks prior to Visit 2 or any intended change during the trial.
* Synovectomy, and/or surgical treatment for RA in the previous 3 months prior to visit 2 or intended indication during the trial.
* Synoviorthesis in the previous 4 weeks prior to Visit 2 or intended indication during the trial.
* Patients in treatment with any other leukotriene inhibitors such as montelukast or zafirlukast 4 weeks prior to Visit 2 or intended use during the trial.
* Initiation of physiotherapy during the 2 weeks before V2, or intended change during the trial
* Patients with history of cardiovascular, renal, neurologic, psychiatric, liver, gastrointestinal (including lactose intolerance ), immunologic or endocrine dysfunction if they are clinically significant.
* Patients with any other known condition or circumstance, which would in the investigator's opinion, prevents compliance or completion of the study
* Patients with history of cancer within the past 5 years, excluding treated basal cell carcinoma
* Patients with chronic infection or acute infections during the 4 weeks before visit 1
* Patients with known positive serology for hepatitis B or C
* Patients with anticoagulant treatment (i.e. dicumarol or derivatives, warfarin)
* Any of the following abnormal laboratory parameters at Visit 2:

  * Impaired hepatic function, defined by serum levels of either Aspartate Aminotransferase (AST)(SGOT), Alanine Aminotransferase (ALT) (SGPT), alkaline phosphatase or bilirubin > 2 x upper limit of normal (ULN)
  * Impaired renal function, defined by serum creatinine > 133 mmol/L (1.5 mg/dl)
  * Hemoglobin values < 10 g/dl
  * White blood cell count <= 3.500 cells/mm3
  * Platelet count of less than 120.000/mm3
  * Severe hypoproteinemia (e.g. in case of severe liver disease or nephrotic syndrome) with albumin < 3.0 g/dl
* Patients with any other abnormal, clinically relevant laboratory values not related to RA
* Patients participating in another clinical trial during the 3 months prior to visit 2
* Previous participation in the randomised period of this study
* Patients with a significant history and/or active alcohol or drug abuse Significant is defined as that which in the opinion of the investigator may either put the patient at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study
* Pregnancy (to be excluded by pregnancy test at visit 1) or breast feeding, and sexually active women with childbearing potential not using a medically approved method of contraception (i.e. oral contraceptives, intrauterine devices, or double-barrier) for at least one month before and throughout the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2001-05; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving 20% improvement assessed by the American College of Rheumatology (ACR) criteria (ACR20) | 3 months

SECONDARY OUTCOMES:
Percentage of patients achieving 50% improvement (ACR50) | 3 months
Number of withdrawals due to lack of efficacy | up to 3 months
Number of swollen joints | up to 3 months
Number of tender joints | up to 3 months
Patient's assessment of pain on a visual analog scale (VAS) | up to 3 months
Patient's global assessment of disease activity by VAS | up to 3 months
Investigator's global assessment of disease activity by VAS | up to 3 months
Patient's assessment of physical function | up to 3 months
  via Health Assessment Questionnaire (HAQ)
Change in erythrocyte sedimentation rate (ESR) | up to 3 months
Change in C-reactive protein (CRP) | up to 3 months
Change in Quality of Life | baseline, 3 months
  assessed by the SF-36 questionnaire
Change in Disease Activity Score (DAS 28) | baseline, up to 3 months
  Disease Activity Score in 28-joint count
Change in duration of morning stiffness | up to 3 months
Consumption of rescue medication | up to 3 months
Number of patients with adverse events | up to 3 months
Number of withdrawals due to adverse events | up to 3 months
Final global assessment of tolerability by investigator on a 4-point scale | 3 months
Patient's assessment of fatigue by VAS | up to 3 months
Number of patients with clinically significant changes in laboratory findings | up to 3 months
Number of patients with clinically significant changes in vital signs | up to 3 months
Number of patients with clinically significant changes in 12-lead ECG | 3 months